CLINICAL TRIAL: NCT03146078
Title: Rate of Progression in USH2A-related Retinal Degeneration
Acronym: RUSH2A
Status: Active, not recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: RUSH2A
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-06

CONDITIONS: Usher Syndrome, Type 2A; Retinitis Pigmentosa 39
MeSH Terms: conditions — Usher syndrome, type 2A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Cohort: Participants with baseline visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and stable fixation and clinically determined [on Octopus 900 Pro] kinetic visual field III4e area 10° or more in the study eye ("primary cohort") will be enrolled into the longitudinal natural history study
- Secondary Cohort: Participants with baseline visual acuity ETDRS letter score of 53 or less [approximate Snellen equivalent 20/100 or worse] or unstable fixation or clinically determined [on Octopus 900 Pro] kinetic visual field III4e area less than 10°in the study eye ("secondary cohort") will be enrolled in the cross-sectional baseline study
- Virtual Reality (VR) Cohort: A subset of sites participating in the VR ancillary study will complete a feasibility questionnaire, including assessment of available space for running the testing procedures. Selected sites will work with VR vendor to complete installation, training, and certification requirements. Eligible participants will be presented with the opportunity to participate in the RUSH2A Extension Study at sites participating in the VR Ancillary Study.
  Participants at VR Sites must consent to the VR Ancillary Study to participate in the RUSH2A Extension Study.

SUMMARY:
The overall goal of this project funded by the Foundation Fighting Blindness is to characterize the natural history of disease progression in patients with USH2A related retinal degeneration associated with congenital hearing loss (Usher syndrome type 2a) or non-syndromic retinitis pigmentosa (RP39).

RUSH2A Extension Study: The purpose of this addendum is to extend RUSH2A to 7- and 9-year visits, with the goal to use longer term data to further develop and support early candidate endpoints as possible clinical trial outcomes.

DETAILED DESCRIPTION:
This natural history study of patients with USH2A mutations will accelerate the development of outcome measures for clinical trials. Sensitive, objective outcome measures of retinal degeneration will greatly facilitate development of treatments for Usher syndrome patients. Together these approaches are expected to have an impact on understanding USH2A-related retinal degeneration, developing experimental treatment protocols, and assessing their effectiveness.

The goals and expected impact of this natural history study are to:

1. Report the natural history of retinal degeneration in patients with biallelic mutations in the USH2A gene
2. Identify sensitive structural and functional outcome measures to use for future multicenter clinical trials in USH2A-related retinal degeneration
3. Identify well-defined subpopulations for future clinical trials of investigative treatments for USH2A-related retinal degeneration

Study Objectives

The primary objectives of the natural history study are to:

1. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the USH2A gene over 4 years, as measured using functional outcome measures (static perimetry, microperimetry, full-field stimulus threshold (FST), electroretinography (ERG), and visual acuity)
2. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the USH2A gene over 4 years, as measured using structural outcome measures (spectral-domain optical coherence tomography (SD-OCT) ellipsoid zone (EZ) area)
3. Investigate structure-function relationships for insights into the mechanisms of retinal degeneration by relating changes in SD-OCT EZ area to visual field progression in individuals with biallelic pathogenic mutations in the USH2A gene
4. Assess for possible genotype, phenotype, and environmental risk factors with progression of the outcome measures at 4 years in individuals with biallelic pathogenic mutations in the USH2A gene

Some additional secondary objectives of this study include:

1. Characterize baseline cross-sectional retinal degeneration associated with biallelic pathogenic mutations in the USH2A gene (as measured using the main outcome measures)
2. Investigate comorbidities associated with disease (baseline cross-sectional) and disease progression (longitudinal natural history study) in individuals with biallelic pathogenic mutations in the USH2A gene
3. Explore patient reported outcome (PRO) measures associated with disease (baseline cross-sectional) and disease progression (longitudinal natural history study) in individuals with biallelic pathogenic mutations in the USH2A gene
4. Evaluate variability and symmetry of left and right eye kinetic perimetry and SD-OCT outcomes at baseline and at 4 years in individuals with biallelic pathogenic mutations in the USH2A gene

RUSH2A Extension Study:

Extension Study Objectives:

Objectives of the RUSH2A Extension Study include evaluating the original study objectives over the longer term (progression on structural and functional outcomes, correlation of progression among outcomes, and factors related to progression) as well as correlating early changes of microperimetry slope, static perimetry slope, full-field stimulus threshold with longer term clinically meaningful outcomes (possible design of early endpoint / late endpoint proposal for FDA). As part of this effort, we are adding virtual reality mobility course testing to RUSH2A as an ancillary study, for a subset of sites, to evaluate its role as a clinically meaningful outcome in future trials.

Virtual Reality (VR) Ancillary Study:

VR Objectives: Specific objectives of VR as part of the RUSH2A Extension Study include:

Correlate early changes of microperimetry, static perimetry, full-field stimulus threshold with longer term clinically meaningful outcomes (possible design of early endpoint / late endpoint proposal for FDA).

Measure changes in progression of disease on VR outcomes, from 7-year to 9-year visit.

Work out logistical issues of multi-center implementation of VR setup and procedures for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to complete the informed consent process
* Ability to return for all study visits over 48 months if in the natural history study
* Age ≥ 8 years
* At least 2 pathogenic or likely pathogenic mutations in USH2A gene from a clinically certified lab report

Ocular Inclusion Criteria

Both eyes must meet all of the following:

* Clinical diagnosis of a rod-cone degeneration
* Clear ocular media and adequate pupil dilation to permit good quality photographic imaging
* Ability to perform kinetic and static perimetry reliably

Exclusion Criteria:

* Mutations in genes that cause autosomal dominant RP, X-linked RP, or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than USH2A
* Expected to enter experimental treatment trial at any time during this study
* History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine)

Ocular Exclusion Criteria

If either eye has any of the following, the patient is not eligible:

* Current vitreous hemorrhage
* Current or any history of rhegmatogenous retinal detachment
* Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia
* History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months
* Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucoma visual field, nerve changes, or glaucoma filtering surgery)
* Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
* Expected to have cataract removal surgery during the study
* History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function
* History of treatment for retinitis pigmentosa that could affect the progression of retinal degeneration (including participation in a clinical trial within the last year or a retained drug delivery device)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential eligibility will be assessed during a routine examination by an investigator prior to obtaining informed consent, as part of usual care
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Characterize Change using Visual Field Sensitivity | Baseline and every year until study completion (4 years)
  Measured by static perimetry with topographic analysis (Hill of Vision)
Characterize Change using Visual Acuity | Baseline and every year until study completion (4 years)
  Best corrected E-ETDRS visual acuity
Characterize Change using Mean Retinal Sensitivity | Baseline and every year until study completion (4 years)
  Measured by fundus-guided microperimetry
Characterize Change in EZ area | Baseline and every year until study completion (4 years)
  Measured by SD-OCT
Characterize Change in Rod- and cone-mediated retinal function | Baseline and every year until study completion (4 years)
  Measured by FST
Characterize Change in Retinal function | Baseline and after four years
  Full-field ERG amplitudes and timing in response to rod- and cone-specific stimuli

SECONDARY OUTCOMES:
MOST-VR Mobility Testing | Seven and nine year visits
  The MOST-VR system measures the locomotion performance of participants who are sighted or visually impaired as they move physically in an empty room and virtually in a maze, under different lighting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jacque Duncan, MD, Study Chair — University of California, San Francisco
Locations (14):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Vitreo-Retinal Associates, Gainesville, Florida
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - OHSU Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Canada
- Centre hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France
- University of Tubingen, Tübingen, Germany
- Radboud University, Nijmegen, Netherlands
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database is available upon request through the public domain on the FFB/Jaeb public website.
Supporting Information: Study Protocol, ICF
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address

REFERENCES:
- See also: public website — http://ffb.jaeb.org

DOCUMENTS (1):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03146078/Prot_001.pdf